CLINICAL TRIAL: NCT00547547
Title: A Phase I Study of a Combination of High Selenium Brassica Juncea With Irinotecan and Capecitabine
Brief Title: High-Selenium Brassica Juncea, Irinotecan, and Capecitabine in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05122; P30CA033572 (NIH); CHNMC-05122; CDR0000570284 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (high-selenium therapy and chemotherapy) (Experimental)
  Interventions: Dietary Supplement: high-selenium Brassica juncea; Drug: capecitabine; Drug: irinotecan hydrochloride

INTERVENTIONS:
Dietary Supplement: high-selenium Brassica juncea — Dose Level A: 3200 mcg orally day -7 through duration of treatment. Dose Level B: 4800 mcg orally day -7 through duration of treatment. Dose Level C: 6400 mcg orally day -7 through duration of treatment. Dose Level D: 7200 mcg orally day -7 through duration of treatment. Dose Level E: 8000 mcg orally day -7 through duration of treatment.
Drug: capecitabine — Dose Level 1: 750 mg/m2, 2x daily x 14 days every 21 days. Dose Level 1.5: 850 mg/m2, 2x daily x 14 days every 21 days. Dose Level 2: 1000 mg/m2, 2x daily x 14 days every 21 days.
Drug: irinotecan hydrochloride — Dose Level 1: 100 mg/m2 on day 1 and day 8 every 21 days. Dose Level -1: 75 mg/m2 on day 1 and day 8 every 21 days.

SUMMARY:
RATIONALE: Brassica juncea that contains high amounts of selenium may slow the growth of cancer cells. Drugs used in chemotherapy, such as irinotecan and capecitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving high-selenium Brassica juncea together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of high-selenium Brassica juncea and capecitabine when given together with irinotecan in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of high-selenium Brassica juncea (BJ-Se) and capecitabine when administered in combination with irinotecan hydrochloride in patients with advanced malignancies.
* To determine the effects of BJ-Se on the pharmacokinetics of irinotecan hydrochloride and capecitabine.

Secondary

* To determine the effect of BJ-Se on the serum selenium and protein profile.
* To correlate response and tolerance to this regimen with expression of key enzymes involved as targets or with the metabolism of the components of treatment, including thymidylate synthase and dihydropyrimidine dehydrogenase.
* To evaluate changes to potential selenium related parameters.

OUTLINE: This is a multicenter, dose-escalation study of high-selenium Brassica juncea (BJ-Se) and capecitabine. The dose of capecitabine is escalated first, followed by dose escalation of BJ-Se.

Patients receive oral BJ-Se on days -7 to 21 in course 1 and on days 1-21 in all other courses. Patients also receive irinotecan IV on days 1 and 8 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.

After the maximum tolerated dose (MTD) of capecitabine and BJ-Se are determined, additional patients are accrued and receive treatment at the MTD. Blood is collected from these patients during course 1 for pharmacokinetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced, biopsy-proven cancer for which there is no standard curative therapy
* Karnofsky Performance status >= 60
* Prior therapy completed at least 3 weeks before protocol treatment initiation with recovery from any side-effects
* Prior capecitabine and/or irinotecan are allowed if subject did not progress while on treatment or within 6 months of treatment with these medications either alone or in combination
* Prior radiation therapy allowed if < 30% of marrow treated
* Alanine aminotransferase (ALT) and alkaline phosphatase with 3x upper limit of normal
* Serum bilirubin within normal limits
* Absolute neutrophil count >= 15000/ul
* Platelet count >= 100,000/ul
* Hemoglobin >= 10 gm/dl - transfusion allowed to achieve this
* Serum creatinine within 1.5 x upper limit of normal
* Ability to understand and sign an IRB approved informed consent
* Ability to use appropriate contraception and no evidence of pregnancy in female patients of reproductive potential

Exclusion Criteria:

* No significant medical or psychiatric condition that would make treatment unsafe
* No active brain metastases (patients who have treated brain metastases and are stable off of steroids are eligible)
* Nursing women
* Patients must be able to comply with protocol related studies and follow-up
* Patients who are UGT1a1 7/7 positive will be excluded from the dose escalation portion of the trial, but may participate in the cohort of patients treated at the MTD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of high-selenium Brassica juncea, irinotecan hydrochloride and capecitabine | After two 21 day cycles of treatment
Toxicity | After two 21 day cycles of treatment
Pharmacokinetics | For patients treated at the MTD only at the end of cycle one of treatment

SECONDARY OUTCOMES:
Serum selenium and protein profile | 21 days after the start of the last cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yun I. Yen, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, Pasadena, California